CLINICAL TRIAL: NCT06072105
Title: Medical Decision Making in Multiple System Atrophy: Developing Personalized Best Medical Care with Integrated Telemedicine and Mobile Palliative Care for Individuals with Multiple System Atrophy
Brief Title: Medical Decision Making in Multiple System Atrophy
Acronym: MeDeMSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Alessandra Fanciulli, Assoc. Prof. MD PhD, Medical University Innsbruck
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1225/2023
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Multiple System Atrophy
Keywords: MSA; Movement disorders; Autonomic dysfunctions; Telemedicine; Palliative care; Caregivers burden
MeSH Terms: conditions — Multiple System Atrophy; Movement Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator): Personalized best medical care.
  Interventions: Other: Multidisciplinary, personalized symptomatic treatment
- Group 2 (Experimental): Personalized best medical care PLUS telemedicine
  Interventions: Other: Telemedicine visits; Other: Multidisciplinary, personalized symptomatic treatment

INTERVENTIONS:
Other: Telemedicine visits — Monthly telemedicine neurological, psychological and neurorehabilitation (physio-, occupational and speech therapy) consultations
  Arms: Group 2
Other: Multidisciplinary, personalized symptomatic treatment — Multidisciplinary, personalized symptomatic treatment plus mobile palliative care interventions (if wished and needed)

SUMMARY:
The goal of this clinical study is to evaluate the effects of a personalized symptomatic treatment plan integrated with monthly telemedicine and mobile palliative care interventions on a population of individuals diagnosed with Multiple System Atrophy (MSA) and their informal caregivers. The aim is to improve the quality of life of MSA patients and their caregivers, as well as provide them with better support during the disease progression.

After a baseline visit, all 46 patients will receive a personalized therapeutic plan (including medical treatment, physiotherapy, logotherapy and occupational therapy excercises and psychological support) and contact with social workers and a palliative care team. They willl then be re-evaluated at 6-,12-, 18- month visits. Semi-structured online interviews at baseline and 12 month visit will collect patients' individual healthcare preferences, which will be taken into account in the preparation of the individual therapeutic plan. Twenty-three patients will be randomized to receive monthly telemedicine visits. Assessment of patients´satisfaction with the therapeutic plan, with the palliative interventions (when they occurred) and the telemedicine visits will be carried over the 18 month period.

Forty-six informal caregivers will be invited to participate with semi-structured online interviews and assessment of their QoL and caregivers' burden.

DETAILED DESCRIPTION:
This is a monocentric, 18-months, randomized, rater-blinded study to evaluate the influence of a multidisciplinary, personalized symptomatic treatment plan with integrated mobile palliative care and telemedicine on the baseline to 18-months change in the QoL of individuals with MSA compared to a sex-, age- and disease-duration matched historical European MSA cohort, whose data is stored at the Medical University of Innsbruck.

We plan to recruit 46 individuals with MSA fulfilling all the inclusionand none of the exclusion criteria. Upon collection of written informed consent, the recruited individuals will be instructed to complete a falls protocol referred to the month preceding the baseline visit, as well as a blood pressure (BP), bladder diary for up to 72 hours prior to the baseline visit. They will subsequently undergo a baseline examination including a comprehensive clinical, psychological and neuro-rehabilitation assessment, as well as an online semi-structured interview aimed at pinpointing the individual therapeutic needs and healthcare preferences. In case additional examinations are needed, these will be carried out on the same day of the baseline visit or, if not possible for individual or appointment reasons, at the earliest possible time point within the given timeframe as outlined in the visit schedule. Upon completion of the baseline visit and examinations, the individualized therapeutic plan, including mobile palliative care offer (for wheelchair-bound individuals) and guidance for self-practiced physio-, speech and occupational exercises will be prepared based on a standardized operational protocol drafted by the study team on the basis of published consensus recommendations, scientific evidence and principles of good clinical practice and adapted to the individual healthcare preferences and therapeutic needs of the recruited individuals.

Six, 12 and 18 months after the baseline visit, in-person visits will be scheduled, including a comprehensive clinical, psychological and neuro-rehabilitation re-assessment of the individual therapeutic needs. Therapeutic adaptations will be made following the standardized operational protocol and adapted to the individual healthcare preferences. In the event that the enrolled subjects are for legitimate reasons unable to travel to hospital, they will be offered the opportunity to complete the scheduled on-site assessments of month 6, 12, and 18 using the CHES online platform.

At month 12 the online semi-structured interview will be repeated to assess for eventual changes in the individual healthcare preferences due to the disease progression.

At month 1, 7 and 13, follow-up phone calls will be scheduled to verify the compliance with the individualized treatment plan and identify barriers to its application.

At month 1, 7, 13 and 18, the study participants will be invited to complete online satisfaction surveys with the overall individualized treatment plan.

Twenty-three patients will be block-wise randomized to receive additional monthly and on-demand neurological, psychological, physio-, occupational and speech therapy (based on individual needs) telemedicine visits through the CHES teleconsultation facility of the Tirol Kliniken.

Upon completion of the telemedicine visit (or on-demand mobile palliative interventions, for wheelchair-bound individuals, whenever needed and wished), brief satisfaction surveys will be sent to the study participants through the CHES platform.

Informal caregivers of the individuals with MSA recruited in the present study will be invited to participate upon written informed consent in an 18 months observational study, with baseline and 12 months semi-structured online interviews and baseline, 6-, 12- and 18 months assessment of their QoL and caregivers' burden.

ELIGIBILITY:
Inclusion Criteria

For individuals with MSA:

* Age ≥30 years at the time of consent;
* Diagnosed with clinically probable or clinically established MSA according to the current MDS MSA criteria (1);
* Life-expectancy of at least 24 months as assessed by the investigator at the time of consent;
* Understands and agrees to comply with the study procedures and provides written informed consent (Note: a legal representative may NOT provide consent on behalf of the subject);
* Signed and dated informed consent document;
* Fluency in German;
* If not able to walk or stand without assistance/support at the time of consent, the participant lives in Tyrol or in another Austrian Region with available mobile palliative care.

For informal caregivers:

* Informal caregiver (i.e. person not receiving payment for his/her caregiving) of an individual with MSA recruited in the present study;
* Life-expectancy of at least 24 months as assessed by the investigator at the time of consent;
* Age≥ 18 years at the time of consent;
* Understands and agrees to provide information as outlined in the study protocol and to engage in semi-structured online interviews;
* Provides signed and dated written informed consent;
* Full legal capacity;
* Fluency in German.

Exclusion Criteria

For individuals with MSA

* Participation in an interventional clinical study at screening and throughout the study that would interfere with the MeDeMSA Care personalized treatment plan or would not permit telemedicine and mobile palliative care strategies;
* Charlson comorbidity index >4 at the time of consent;
* Other major underlying medical conditions that may confound interpretation of study results as assessed by the investigator.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in the EQ-5D-5L score | Baseline to 18-months
  European Quality of life - 5 Dimensions - 5 Levels. This is a 5 dimensions assessment of mobility, self-care, usual activities, pain/discomfort and anxiety/depression that provides a single summary index value for health status. It also includes the EQ-VAS, a self-rating of overall health on a visual analogue scale (VAS), ranging from 0 (worst imaginable health state) to 100 (best imaginable health state). A summary index with a maximum score of 1 can be derived from the five dimensions of EQ-5D by conversion with a table of scores. The maximum score of 1 indicates the best health state, in contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems.

SECONDARY OUTCOMES:
Changes in the MSA-QoL score and subscores | Baseline to 6-, 12- and 18-months
  The Multiple System Atrophy - Quality of Life,is a questionnaire composed of 40 items investigating several MSA-specific motor and non-motor symptoms, as well as their perceived impact on daily life and a numeric rating scale to assess the QoL of individuals diagnosed with MSA. Scores on each of the subscales of the MSA are derived by summing the respective items and transforming to a range of 0-100, with higher scores on each scale indicating a higher impact of the disease on the aspect measured by each subscale.
Change in motor and non-motor scales | Baseline to 6-, 12- and 18-months
  It includes total and subscores, as video-based, rater-blinded assessment of the UMSARS (Unified Multiple System Atrophy Rating Scale) motor score and Hoehn & Yahr changes over the study period. In both the scales a higher score is related to a higher impact of the disease on the aspect measured.
Time to clinical milestones | over the 18-months study period
  The clinical milestones are falls at least once a day, feeding by nasogastric tube or gastrostomy, unintelligible speech, indwelling catheter, wheelchair dependency.
Changes in the individual healthcare preferences assessed by means of the Autonomy Preference Index (API) | Baseline to 12- months
  Assessment of individual preferences about the individual healthcare
In-person and telemedicine medical, psychological and neurorehabilitation interventional needs of individuals with MSA | over the 18-months study period
  Registration of the need of support required by MSA patients
Change in the Short Assessment of Patient Satisfaction (SAPS) referred to the overall individualized treatment plan | Month 1 to 7, 13 and 18
  Assessment of patients´ level of satisfaction with the individuaized treatment plan
Individual satisfaction with the single telemedicine and mobile palliative interventions | over the 18-months study period
  The individual satisfaction will be assessed by means of online numeric rating scales and open-ended questions
Healthcare professionals satisfaction with the single telemedicine and mobile palliative interventions | over the 18-months study period
  The individual healthcare professionals satisfaction will be assessed by means of online numeric rating scales and open-ended questions
Number of medical complications | over the 18-months study period
  Record of number of medical complications occurred (e.g. falls with or w/o injuries, urinary tract infections, choking, aspiration pneumonia, hospitalizations, death, others)
Single-intervention and cumulative healthcare costs | over the 18-months study period
  Record of healthcare costs
Changes in the EQ-5D-5L score of informal caregivers of individuals with MSA recruited in the present study | Baseline to 6-, 12- and 18-months
  European Quality of life - 5 Dimensions - 5 Levels. This is a 5 dimensions assessment of mobility, self-care, usual activities, pain/discomfort and anxiety/depression that provides a single summary index value for health status. It also includes the EQ-VAS, a self-rating of overall health on a visual analogue scale (VAS), ranging from 0 (worst imaginable health state) to 100 (best imaginable health state). A summary index with a maximum score of 1 can be derived from the five dimensions of EQ-5D by conversion with a table of scores. The maximum score of 1 indicates the best health state, in contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems.
Change in the Carers quality-of-life questionnaire for parkinsonism (PQoL Carers) score and other caregiver-burden indicators in informal caregivers of individuals with MSA recruited in the present study | Baseline to 6-, 12- and 18-months
  The Parkinsonism Carers Quality of Life, is a questionnaire composed of 26 items and is a concise instrument with adequate psychometric qualities to assess the QoL of the caregivers of people with atypical Parkinsonism. A score of 0 indicates the best level of QoL, whereas a score of 100 the worst level.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Fanciulli, MD PhD, Principal Investigator — Medizinische Universität Innsbruck
Locations (1):
- Innsbruck Medical University, Innsbruck, Austria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wenning GK, Stankovic I, Vignatelli L, Fanciulli A, Calandra-Buonaura G, Seppi K, Palma JA, Meissner WG, Krismer F, Berg D, Cortelli P, Freeman R, Halliday G, Hoglinger G, Lang A, Ling H, Litvan I, Low P, Miki Y, Panicker J, Pellecchia MT, Quinn N, Sakakibara R, Stamelou M, Tolosa E, Tsuji S, Warner T, Poewe W, Kaufmann H. The Movement Disorder Society Criteria for the Diagnosis of Multiple System Atrophy. Mov Disord. 2022 Jun;37(6):1131-1148. doi: 10.1002/mds.29005. Epub 2022 Apr 21. PMID 35445419
- [Background] Wenning GK, Krismer F. Multiple system atrophy. Handb Clin Neurol. 2013;117:229-41. doi: 10.1016/B978-0-444-53491-0.00019-5. PMID 24095129
- [Background] Kwakkenbos L, Fransen J, Vonk MC, Becker ES, Jeurissen M, van den Hoogen FH, van den Ende CH. A comparison of the measurement properties and estimation of minimal important differences of the EQ-5D and SF-6D utility measures in patients with systemic sclerosis. Clin Exp Rheumatol. 2013 Mar-Apr;31(2 Suppl 76):50-6. Epub 2013 Jul 22. PMID 23910610
- [Background] Fanciulli A, Wenning GK. Multiple-system atrophy. N Engl J Med. 2015 Jan 15;372(3):249-63. doi: 10.1056/NEJMra1311488. No abstract available. PMID 25587949
- [Background] Cortelli P, Calandra-Buonaura G, Benarroch EE, Giannini G, Iranzo A, Low PA, Martinelli P, Provini F, Quinn N, Tolosa E, Wenning GK, Abbruzzese G, Bower P, Alfonsi E, Ghorayeb I, Ozawa T, Pacchetti C, Pozzi NG, Vicini C, Antonini A, Bhatia KP, Bonavita J, Kaufmann H, Pellecchia MT, Pizzorni N, Schindler A, Tison F, Vignatelli L, Meissner WG. Stridor in multiple system atrophy: Consensus statement on diagnosis, prognosis, and treatment. Neurology. 2019 Oct 1;93(14):630-639. doi: 10.1212/WNL.0000000000008208. PMID 31570638
- [Background] Calandra-Buonaura G, Alfonsi E, Vignatelli L, Benarroch EE, Giannini G, Iranzo A, Low PA, Martinelli P, Provini F, Quinn N, Tolosa E, Wenning GK, Abbruzzese G, Bower P, Antonini A, Bhatia KP, Bonavita J, Pellecchia MT, Pizzorni N, Tison F, Ghorayeb I, Meissner WG, Ozawa T, Pacchetti C, Pozzi NG, Vicini C, Schindler A, Cortelli P, Kaufmann H. Dysphagia in multiple system atrophy consensus statement on diagnosis, prognosis and treatment. Parkinsonism Relat Disord. 2021 May;86:124-132. doi: 10.1016/j.parkreldis.2021.03.027. Epub 2021 Mar 30. PMID 33839029
- [Background] Brignole M, Moya A, de Lange FJ, Deharo JC, Elliott PM, Fanciulli A, Fedorowski A, Furlan R, Kenny RA, Martin A, Probst V, Reed MJ, Rice CP, Sutton R, Ungar A, van Dijk JG; ESC Scientific Document Group. 2018 ESC Guidelines for the diagnosis and management of syncope. Eur Heart J. 2018 Jun 1;39(21):1883-1948. doi: 10.1093/eurheartj/ehy037. No abstract available. PMID 29562304
- [Background] Gibbons CH, Schmidt P, Biaggioni I, Frazier-Mills C, Freeman R, Isaacson S, Karabin B, Kuritzky L, Lew M, Low P, Mehdirad A, Raj SR, Vernino S, Kaufmann H. The recommendations of a consensus panel for the screening, diagnosis, and treatment of neurogenic orthostatic hypotension and associated supine hypertension. J Neurol. 2017 Aug;264(8):1567-1582. doi: 10.1007/s00415-016-8375-x. Epub 2017 Jan 3. PMID 28050656
- [Background] Groen J, Pannek J, Castro Diaz D, Del Popolo G, Gross T, Hamid R, Karsenty G, Kessler TM, Schneider M, 't Hoen L, Blok B. Summary of European Association of Urology (EAU) Guidelines on Neuro-Urology. Eur Urol. 2016 Feb;69(2):324-33. doi: 10.1016/j.eururo.2015.07.071. Epub 2015 Aug 22. PMID 26304502
- [Background] Jordan J, Fanciulli A, Tank J, Calandra-Buonaura G, Cheshire WP, Cortelli P, Eschlboeck S, Grassi G, Hilz MJ, Kaufmann H, Lahrmann H, Mancia G, Mayer G, Norcliffe-Kaufmann L, Pavy-Le Traon A, Raj SR, Robertson D, Rocha I, Reuter H, Struhal W, Thijs RD, Tsioufis KP, Gert van Dijk J, Wenning GK, Biaggioni I. Management of supine hypertension in patients with neurogenic orthostatic hypotension: scientific statement of the American Autonomic Society, European Federation of Autonomic Societies, and the European Society of Hypertension. J Hypertens. 2019 Aug;37(8):1541-1546. doi: 10.1097/HJH.0000000000002078. PMID 30882602
- [Background] Randerath W, Verbraecken J, Andreas S, Arzt M, Bloch KE, Brack T, Buyse B, De Backer W, Eckert DJ, Grote L, Hagmeyer L, Hedner J, Jennum P, La Rovere MT, Miltz C, McNicholas WT, Montserrat J, Naughton M, Pepin JL, Pevernagie D, Sanner B, Testelmans D, Tonia T, Vrijsen B, Wijkstra P, Levy P. Definition, discrimination, diagnosis and treatment of central breathing disturbances during sleep. Eur Respir J. 2017 Jan 18;49(1):1600959. doi: 10.1183/13993003.00959-2016. Print 2017 Jan. PMID 27920092
- [Background] Jasemi M, Valizadeh L, Zamanzadeh V, Keogh B. A Concept Analysis of Holistic Care by Hybrid Model. Indian J Palliat Care. 2017 Jan-Mar;23(1):71-80. doi: 10.4103/0973-1075.197960. PMID 28216867
- [Background] Hepgul N, Wilson R, Yi D, Evans C, Bajwah S, Crosby V, Wilcock A, Lindsay F, Byrne A, Young C, Groves K, Smith C, Burman R, Chaudhuri KR, Silber E, Higginson IJ, Gao W. Immediate versus delayed short-term integrated palliative care for advanced long-term neurological conditions: the OPTCARE Neuro RCT. Southampton (UK): NIHR Journals Library; 2020 Sep. Available from http://www.ncbi.nlm.nih.gov/books/NBK561537/ PMID 32902934
- [Background] van Vliet LM, Gao W, DiFrancesco D, Crosby V, Wilcock A, Byrne A, Al-Chalabi A, Chaudhuri KR, Evans C, Silber E, Young C, Malik F, Quibell R, Higginson IJ; OPTCARE Neuro. How integrated are neurology and palliative care services? Results of a multicentre mapping exercise. BMC Neurol. 2016 May 10;16:63. doi: 10.1186/s12883-016-0583-6. PMID 27165157
- [Background] Adams JL, Myers TL, Waddell EM, Spear KL, Schneider RB. Telemedicine: A valuable tool in neurodegenerative diseases. Curr Geriatr Rep. 2020 Jun;9(2):72-81. doi: 10.1007/s13670-020-00311-z. Epub 2020 Mar 14. PMID 32509504
- [Background] Borders JC, Sevitz JS, Malandraki JB, Malandraki GA, Troche MS. Objective and Subjective Clinical Swallowing Outcomes via Telehealth: Reliability in Outpatient Clinical Practice. Am J Speech Lang Pathol. 2021 Mar 26;30(2):598-608. doi: 10.1044/2020_AJSLP-20-00234. Epub 2021 Feb 8. PMID 33555954
- [Background] Morris ME, Slade SC, Wittwer JE, Blackberry I, Haines S, Hackney ME, McConvey VB. Online Dance Therapy for People With Parkinson's Disease: Feasibility and Impact on Consumer Engagement. Neurorehabil Neural Repair. 2021 Dec;35(12):1076-1087. doi: 10.1177/15459683211046254. Epub 2021 Sep 29. PMID 34587834
- [Background] Tamplin J, Morris ME, Baker FA, Sousa TV, Haines S, Dunn S, Tull V, Vogel AP. ParkinSong Online: protocol for a telehealth feasibility study of therapeutic group singing for people with Parkinson's disease. BMJ Open. 2021 Dec 20;11(12):e058953. doi: 10.1136/bmjopen-2021-058953. PMID 34930750
- [Background] Vellata C, Belli S, Balsamo F, Giordano A, Colombo R, Maggioni G. Effectiveness of Telerehabilitation on Motor Impairments, Non-motor Symptoms and Compliance in Patients With Parkinson's Disease: A Systematic Review. Front Neurol. 2021 Aug 26;12:627999. doi: 10.3389/fneur.2021.627999. eCollection 2021. PMID 34512495
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Background] Miyashita M, Narita Y, Sakamoto A, Kawada N, Akiyama M, Kayama M, Suzukamo Y, Fukuhara S. Care burden and depression in caregivers caring for patients with intractable neurological diseases at home in Japan. J Neurol Sci. 2009 Jan 15;276(1-2):148-52. doi: 10.1016/j.jns.2008.09.022. Epub 2008 Oct 26. PMID 18954877
- [Background] Wiblin L, Lee M, Burn D. Palliative care and its emerging role in Multiple System Atrophy and Progressive Supranuclear Palsy. Parkinsonism Relat Disord. 2017 Jan;34:7-14. doi: 10.1016/j.parkreldis.2016.10.013. Epub 2016 Oct 19. PMID 28341224
- [Background] Gallop K, Pham N, Maclaine G, Saunders E, Black B, Hubig L, Acaster S. Health-related quality-of-life and burden for caregivers of individuals with neurogenic orthostatic hypotension. Neurodegener Dis Manag. 2023 Feb;13(1):35-45. doi: 10.2217/nmt-2022-0015. Epub 2022 Nov 16. PMID 36382590
- [Background] Dayal AM, Jenkins ME, Jog MS, Kimpinski K, MacDonald P, Gofton TE. Palliative Care Discussions in Multiple System Atrophy: A Retrospective Review. Can J Neurol Sci. 2017 May;44(3):276-282. doi: 10.1017/cjn.2016.439. Epub 2017 Feb 7. PMID 28166857
- [Background] Strupp J, Kunde A, Galushko M, Voltz R, Golla H. Severely Affected by Parkinson Disease: The Patient's View and Implications for Palliative Care. Am J Hosp Palliat Care. 2018 Apr;35(4):579-585. doi: 10.1177/1049909117722006. Epub 2017 Jul 26. PMID 28743187
- [Background] Wiblin L, Durcan R, Lee M, Brittain K. The Importance of Connection to Others in QoL in MSA and PSP. Parkinsons Dis. 2017;2017:5283259. doi: 10.1155/2017/5283259. Epub 2017 Sep 28. PMID 29093980
- [Background] Bloem BR, Henderson EJ, Dorsey ER, Okun MS, Okubadejo N, Chan P, Andrejack J, Darweesh SKL, Munneke M. Integrated and patient-centred management of Parkinson's disease: a network model for reshaping chronic neurological care. Lancet Neurol. 2020 Jul;19(7):623-634. doi: 10.1016/S1474-4422(20)30064-8. Epub 2020 May 25. PMID 32464101
- [Background] Pinto S, Caldeira S, Martins JC. e-Health in palliative care: review of literature, Google Play and App Store. Int J Palliat Nurs. 2017 Aug 2;23(8):394-401. doi: 10.12968/ijpn.2017.23.8.394. PMID 28854054
- [Background] Chan LML, Yan OY, Lee JJJ, Lam WWT, Lin CC, Auyeung M, Bloem BR, Kwok JYY. Effects of Palliative Care for Progressive Neurologic Diseases: A Systematic Review and Meta-Analysis. J Am Med Dir Assoc. 2023 Feb;24(2):171-184. doi: 10.1016/j.jamda.2022.11.001. Epub 2022 Dec 5. PMID 36481217
- [Background] Coon EA, Golden EP, Bryarly M, McGregor T, Nguyen BN, Moutvic MA, Cutsforth-Gregory JK, Stevens PM, Chou CZ, Rhee L, Vernino S. A call for multiple system atrophy centers of excellence. Clin Auton Res. 2022 Jun;32(3):205-208. doi: 10.1007/s10286-022-00866-1. Epub 2022 May 12. No abstract available. PMID 35552950
- [Background] Pillas M, Selai C, Quinn NP, Lees A, Litvan I, Lang A, Bower J, Burn D, Low P, Schrag A. Development and validation of a carers quality-of-life questionnaire for parkinsonism (PQoL Carers). Qual Life Res. 2016 Jan;25(1):81-8. doi: 10.1007/s11136-015-1071-y. Epub 2015 Aug 12. PMID 26264781
- [Background] Schrag A, Selai C, Jahanshahi M, Quinn NP. The EQ-5D--a generic quality of life measure-is a useful instrument to measure quality of life in patients with Parkinson's disease. J Neurol Neurosurg Psychiatry. 2000 Jul;69(1):67-73. doi: 10.1136/jnnp.69.1.67. PMID 10864606
- [Background] Schrag A, Selai C, Mathias C, Low P, Hobart J, Brady N, Quinn NP. Measuring health-related quality of life in MSA: the MSA-QoL. Mov Disord. 2007 Dec;22(16):2332-8. doi: 10.1002/mds.21649. PMID 17914730
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Sletten DM, Suarez GA, Low PA, Mandrekar J, Singer W. COMPASS 31: a refined and abbreviated Composite Autonomic Symptom Score. Mayo Clin Proc. 2012 Dec;87(12):1196-201. doi: 10.1016/j.mayocp.2012.10.013. PMID 23218087
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Frauscher B, Ehrmann L, Zamarian L, Auer F, Mitterling T, Gabelia D, Brandauer E, Delazer M, Poewe W, Hogl B. Validation of the Innsbruck REM sleep behavior disorder inventory. Mov Disord. 2012 Nov;27(13):1673-8. doi: 10.1002/mds.25223. PMID 23192924
- [Background] Chung F, Yegneswaran B, Liao P, Chung SA, Vairavanathan S, Islam S, Khajehdehi A, Shapiro CM. STOP questionnaire: a tool to screen patients for obstructive sleep apnea. Anesthesiology. 2008 May;108(5):812-21. doi: 10.1097/ALN.0b013e31816d83e4. PMID 18431116
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Freynhagen R, Baron R, Gockel U, Tolle TR. painDETECT: a new screening questionnaire to identify neuropathic components in patients with back pain. Curr Med Res Opin. 2006 Oct;22(10):1911-20. doi: 10.1185/030079906X132488. PMID 17022849
- [Background] Wenning GK, Tison F, Seppi K, Sampaio C, Diem A, Yekhlef F, Ghorayeb I, Ory F, Galitzky M, Scaravilli T, Bozi M, Colosimo C, Gilman S, Shults CW, Quinn NP, Rascol O, Poewe W; Multiple System Atrophy Study Group. Development and validation of the Unified Multiple System Atrophy Rating Scale (UMSARS). Mov Disord. 2004 Dec;19(12):1391-402. doi: 10.1002/mds.20255. PMID 15452868
- [Background] Ende J, Kazis L, Ash A, Moskowitz MA. Measuring patients' desire for autonomy: decision making and information-seeking preferences among medical patients. J Gen Intern Med. 1989 Jan-Feb;4(1):23-30. doi: 10.1007/BF02596485. PMID 2644407
- [Background] Dillen K, Goereci Y, Dunkl V, Muller A, Fink GR, Voltz R, Hocaoglu M, Warnke C, Golla H. Cultural adaptation of the Integrated Palliative care Outcome Scale for neurological symptoms. Palliat Support Care. 2023 Dec;21(6):1059-1068. doi: 10.1017/S1478951523000238. PMID 37039454
- [Background] Hawthorne G, Sansoni J, Hayes L, Marosszeky N, Sansoni E. Measuring patient satisfaction with health care treatment using the Short Assessment of Patient Satisfaction measure delivered superior and robust satisfaction estimates. J Clin Epidemiol. 2014 May;67(5):527-37. doi: 10.1016/j.jclinepi.2013.12.010. PMID 24698296
- [Background] da Silva BA, Faria CDCM, Santos MP, Swarowsky A. Assessing Timed Up and Go in Parkinson's disease: Reliability and validity of Timed Up and Go Assessment of biomechanical strategies. J Rehabil Med. 2017 Nov 21;49(9):723-731. doi: 10.2340/16501977-2254. PMID 28951938
- [Background] Lang JT, Kassan TO, Devaney LL, Colon-Semenza C, Joseph MF. Test-Retest Reliability and Minimal Detectable Change for the 10-Meter Walk Test in Older Adults With Parkinson's disease. J Geriatr Phys Ther. 2016 Oct-Dec;39(4):165-70. doi: 10.1519/JPT.0000000000000068. PMID 26428902
- [Background] Perez-Lloret S, van de Warrenburg B, Rossi M, Rodriguez-Blazquez C, Zesiewicz T, Saute JAM, Durr A, Nishizawa M, Martinez-Martin P, Stebbins GT, Schrag A, Skorvanek M; members of the MDS Rating Scales Review Committee. Assessment of Ataxia Rating Scales and Cerebellar Functional Tests: Critique and Recommendations. Mov Disord. 2021 Feb;36(2):283-297. doi: 10.1002/mds.28313. Epub 2020 Oct 6. PMID 33022077
- [Background] Alonso CCG, de Freitas PB, Pires RS, De Oliveira DL, Freitas SMSF. Exploring the ability of strength and dexterity tests to detect hand function impairment in individuals with Parkinson's disease. Physiother Theory Pract. 2023 Feb;39(2):395-404. doi: 10.1080/09593985.2021.2013371. Epub 2021 Dec 12. PMID 34895020
- [Background] Ona ED, Jardon A, Cuesta-Gomez A, Sanchez-Herrera-Baeza P, Cano-de-la-Cuerda R, Balaguer C. Validity of a Fully-Immersive VR-Based Version of the Box and Blocks Test for Upper Limb Function Assessment in Parkinson's Disease. Sensors (Basel). 2020 May 13;20(10):2773. doi: 10.3390/s20102773. PMID 32414177
- [Background] De Dobbeleer L, Beyer I, Hansen AM, Molbo D, Mortensen EL, Lund R, Bautmans I. Grip Work Measurement with the Jamar Dynamometer: Validation of a Simple Equation for Clinical Use. J Nutr Health Aging. 2019;23(2):221-224. doi: 10.1007/s12603-019-1155-4. PMID 30697635
- [Background] Bartolome G, Starrost U, Schroter-Morasch H, Schilling B, Fischbacher L, Kues L, Graf S, Ziegler W. Validation of the Munich Swallowing Score (MUCSS) in patients with neurogenic dysphagia: A preliminary study. NeuroRehabilitation. 2021;49(3):445-457. doi: 10.3233/NRE-210011. PMID 34180423
- [Background] Eschlbock S, Wenning G, Fanciulli A. Evidence-based treatment of neurogenic orthostatic hypotension and related symptoms. J Neural Transm (Vienna). 2017 Dec;124(12):1567-1605. doi: 10.1007/s00702-017-1791-y. Epub 2017 Oct 22. PMID 29058089
- [Background] Wenning GK, Geser F, Krismer F, Seppi K, Duerr S, Boesch S, Kollensperger M, Goebel G, Pfeiffer KP, Barone P, Pellecchia MT, Quinn NP, Koukouni V, Fowler CJ, Schrag A, Mathias CJ, Giladi N, Gurevich T, Dupont E, Ostergaard K, Nilsson CF, Widner H, Oertel W, Eggert KM, Albanese A, del Sorbo F, Tolosa E, Cardozo A, Deuschl G, Hellriegel H, Klockgether T, Dodel R, Sampaio C, Coelho M, Djaldetti R, Melamed E, Gasser T, Kamm C, Meco G, Colosimo C, Rascol O, Meissner WG, Tison F, Poewe W; European Multiple System Atrophy Study Group. The natural history of multiple system atrophy: a prospective European cohort study. Lancet Neurol. 2013 Mar;12(3):264-74. doi: 10.1016/S1474-4422(12)70327-7. Epub 2013 Feb 5. PMID 23391524
- [Background] Siebert U, Alagoz O, Bayoumi AM, Jahn B, Owens DK, Cohen DJ, Kuntz KM. State-transition modeling: a report of the ISPOR-SMDM Modeling Good Research Practices Task Force-3. Med Decis Making. 2012 Sep-Oct;32(5):690-700. doi: 10.1177/0272989X12455463. PMID 22990084
- [Background] Drummond MF, Schwartz JS, Jonsson B, Luce BR, Neumann PJ, Siebert U, Sullivan SD. Key principles for the improved conduct of health technology assessments for resource allocation decisions. Int J Technol Assess Health Care. 2008 Summer;24(3):244-58; discussion 362-8. doi: 10.1017/S0266462308080343. PMID 18601792